CLINICAL TRIAL: NCT01025453
Title: Phase II Study Evaluating the Combination of Temsirolimus and Sorafenib in the Treatment of Radioactive Iodine Refractory Thyroid Cancer
Brief Title: Combination of Temsirolimus and Sorafenib in the Treatment of Radioactive Iodine Refractory Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-148
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Thyroid Cancer
Keywords: thyroid; follicular cell; papillary cell; Hurthle cell; BAY 43-9006; Temsirolimus; Sorafenib; 09-148
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Diseases | interventions — temsirolimus; Sorafenib

ARMS (1):
- Pts getting Temsirolimus and Sorafenib (Experimental): We propose a phase II study to evaluate the efficacy of the combination sorafenib with temsirolimus in patients with thyroid cancer of follicular cell origin (e.g., papillary, follicular, Hurthle cell). A maximum of 36 subjects will be evaluated during the study. Restaging scans, with evaluation of response, will be done every 2 cycles (8 weeks of treatment). Treatment will continue until clinical disease progression, unacceptable toxicity, treatment delay > 4 weeks, or at the discretion of the treating physician or patient.
  Interventions: Drug: Temsirolimus and Sorafenib

INTERVENTIONS:
Drug: Temsirolimus and Sorafenib — Treatment will be with sorafenib 200 mg orally twice a day and temsirolimus 25 mg intravenous weekly. A cycle will be equivalent to 4 weeks of treatment.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, the combination of sorafenib and temsirolimus will have on thyroid cancer. Treatment guidelines from the National Comprehensive Cancer Network include sorafenib as a treatment option for thyroid cancer.

Temsirolimus is an intravenous medication that is FDA approved for other type of cancers. In laboratory studies, the addition of temsirolimus to sorafenib works better than sorafenib alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histopathologically confirmed at MSKCC thyroid carcinoma of follicular cell origin (D-TC-FCO), which includes papillary, follicular, Hürthle cell histology, or anaplastic along with their respective variants.
* Available pathology for RAF mutational testing (e.g., paraffin block or 5-10 unstained slides). It is not required that mutational testing be completed before starting the clinical study.
* Patients must have surgically inoperable and/or recurrent/metastatic disease.
* Patients must have a PET scan prior to the protocol start date and have at least one FDGavid lesion that has not been removed surgically or radiated (unless it has progressed by RECIST criteria after the completion of radiation therapy and is still FDG-avid). FDGavidity will be defined as any focus of increased FDG uptake greater than normal activity with SUV maximum levels greater than or equal to 3. PET scan can have been done at any time prior to the start of therapy, although it is recommended that it be done within 3 months prior to the start of therapy.
* Patients must have measurable disease by RECIST criteria, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan; performed ≤ 4 weeks of protocol start date.
* Patients must have progressive disease defined by at least one of the following occurring during or after previous treatment (including RAI treatment):
* The presence of new or progressive lesions on CT/MRI.
* New lesions on bone scan or PET scan.
* Rising thyroglobulin level (documented by a minimum of three consecutive rises, with an interval of > 1 week between each determination).
* Prior RAI therapy is allowed if > 3 months prior to initiation of therapy on this protocol and evidence of progression (as defined above) has been documented in the interim. A diagnostic study using <10 mCi of RAI is not considered RAI therapy.
* Patients may have received prior external beam radiation therapy to index lesions ≥ 4 weeks prior to initiation of therapy on this protocol if there has been documented progression by RECIST criteria. Prior external beam radiation therapy to the non-index lesions is allowed if ≥ 4 weeks prior to initiation of therapy on this protocol.
* ECOG performance status ≤ 2 (or Karnofsky performance status ≥ 60%).
* Patients must have normal organ and marrow function as defined below:
* Absolute neutrophil count ≥1,500/mcL
* Platelets ≥100,000/mcL
* Total bilirubin ≤ 1.5 X institutional ULN
* AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional ULN
* Creatinine ≤ 1.5 X institutional ULN OR
* Creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above 1.5 X institutional ULN [in this circumstance, either of a measured level based on a 24 hour urine collection, or a calculated level using the Cockcroft and Gault equation: (140 - age in years) X (weight in kg) X (0.85 if female)/72 X serum Cr may be used].
* International normalized ratio (INR) ≤ 1.5 (or in range INR, usually between 2 and 3, if patient is on a stable dose of therapeutic warfarin).
* *ULN = upper limit of normal
* **unless liver metastasis present in which AST/ALT should be < 5 x ULN.
* Ability to understand and the willingness to sign a written informed consent document.
* Age 21 years old or older.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Patients with known history of active intraparenchymal brain metastasis within previous 3 months.
* Serious or non-healing wound, ulcer, or bone fracture.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment.
* Patients with a reported history of clinically active diverticulosis or diverticulitis in the prior 3 years.
* Patients with clinically significant cardiovascular disease as defined by the following:
* History of CVA within past 6 months
* Myocardial infarction, CABG or unstable angina within past 6 months
* New York Heart Association grade III or greater congestive heart failure or Canadian Cardiovascular Class grade III or greater angina within past 6 months (Appendices B&C) Clinically significant peripheral vascular disease within past 6 months
* Pulmonary embolism, DVT, or other thromboembolic event within past 6 months
* Uncontrolled coronary artery disease, angina, congestive heart failure, or ventricular arrhythmia requiring acute medical management within past 6 months
* History of myocardial infarct, cerebrovascular accident, or transient ischemic event within the past 6 month
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* While the use of Angiotensin-Converting Enzyme (ACE) inhibitors is not absolutely excluded, efforts should be made to see if patients on ACE inhibitors can be taken off the medication or switched to another medication.
* Pregnant women will be ineligible; breastfeeding should be discontinued if the mother is treated with study drugs.
* The use of agents that inhibit or induce CYP3A metabolism is not strictly prohibited, but should be avoided if possible. Potential CYP3A inducing agents include carbamazepine, phenytoin, barbiturates, rifabutin, rifampicin, and St. John's Wort. Potential CYP3A inhibitors include protease inhibitors, antifungals, macrolide antibiotics, nefazodone, and selective serotonin inhibitors.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-12-01 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sherman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pts Getting Temsirolimus and Sorafenib
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pts Getting Temsirolimus and Sorafenib
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 64 [30 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 25
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Reponse Rate of the Combination Sorafenib and Temsirolimus in I-131 Refractory Thyroid Cancer.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 2 years
Population: 7 participants were not evaluable because they came off treatment before the first radiographic scan for reasons other than progression of disease, including but not limited to excessive toxicity (n=1), withdrawal of consent (n=3), and seeing other treatment (n=1).
Measure: Count of Participants; unit: Participants
Arm/Group | Pts Getting Temsirolimus and Sorafenib
Number analyzed (Participants) | 30
Participants
  Partial Response | 8
  Stable Disease | 21
  Disease Progression | 1

2. Secondary Outcome: Duration of Study Treatment for Participants With and Without BRAF Mutations
Time Frame: 6 years
Population: The analysis separated the participants into 2 groups (number of patients with BRAF V600E Mutation and number of patients without BRAF V600E Mutation)
Measure: Median (Full Range); unit: months
Arm/Group | Pts Getting Temsirolimus and Sorafenib
Number analyzed (Participants) | 36
months
  Pts with BRAF V600E Mutation: number analyzed (Participants) | 10
  Pts with BRAF V600E Mutation | 5.2 [0.7 to 63]
  Pts w/o BRAF V600E Mutation: number analyzed (Participants) | 26
  Pts w/o BRAF V600E Mutation | 6.7 [0.5 to 25.6]

3. Secondary Outcome: Percentage of Participants With Progression-free Survival Under the Combination Sorafenib and Temsirolimus in I-131 Refractory Thyroid Cancer.
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 1 year
Measure: Number; unit: percentage of patients
Arm/Group | Pts Getting Temsirolimus and Sorafenib
Number analyzed (Participants) | 37
percentage of patients | 30.5

4. Secondary Outcome: Safety and Tolerability for the Combination Sorafenib and Temsirolimus in I-131 Refractory Thyroid Cancer.
Description: Participant toxicities evaluated by CTCAE version 4.0
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Pts Getting Temsirolimus and Sorafenib
Number analyzed (Participants) | 37
Participants | 37

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Pts Getting Temsirolimus and Sorafenib
All-Cause Mortality (participants affected / at risk) | 32/37
Serious Adverse Events (participants affected / at risk) | 23/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pts Getting Temsirolimus and Sorafenib (N=37)
Abdominal Pain (Gastrointestinal disorders) | 3
Alanine aminotransferase increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 1
Appendicitis (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 5
Catheter related infection (Infections and infestations) | 2
Chest pain - cardiac (Cardiac disorders) | 1
Colonic perforation (Gastrointestinal disorders) | 2
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (General disorders) | 1
Creatinine increased (Investigations) | 1
Death NOS (General disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 3
Delirium (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 2
Fever (General disorders) | 3
Headache (Nervous system disorders) | 1
Heart failure (Cardiac disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypertension (Vascular disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Lung infection (Infections and infestations) | 2
Lymphocyte count decreased (Investigations) | 1
Mediastinal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Non-cardiac chest pain (General disorders) | 3
Oral pain (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Paresthesia (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Sudden death NOS (General disorders) | 1
Thromboembolic event (Vascular disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Urinary tract infection (Infections and infestations) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Wound infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pts Getting Temsirolimus and Sorafenib (N=37)
Hyperglycemia (Metabolism and nutrition disorders) | 21
Platelet count decreased (Investigations) | 11
Fatigue (General disorders) | 14
Aspartate aminotransferase increased (Investigations) | 6
Diarrhea (Gastrointestinal disorders) | 11
Alanine aminotransferase increased (Investigations) | 8
Hypertriglyceridemia (Metabolism and nutrition disorders) | 6
Nausea (Gastrointestinal disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 12
Hypertension (Vascular disorders) | 15
Mucositis oral (Gastrointestinal disorders) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6
Anemia (Blood and lymphatic system disorders) | 7
Weight loss (Investigations) | 7
White blood cell decreased (Investigations) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Dysphagia (Gastrointestinal disorders) | 5
Headache (Nervous system disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Edema limbs (General disorders) | 4
Fever (General disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Oral pain (Gastrointestinal disorders) | 2
Creatinine increased (Investigations) | 2
Non-cardiac chest pain (General disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Sinus tachycardia (Cardiac disorders) | 2
Colonic perforation (Gastrointestinal disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT01025453/Prot_SAP_000.pdf